CLINICAL TRIAL: NCT05780411
Title: A Comprehensive Study of Cancer Survivor Syndrome in Adult Egyptian Patients With Hematological Neoplasms
Brief Title: Cancer Survivorship in Hematologic Malignancies
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Roaa Mohammed Mohammed Saleh, Resident Physician, Assiut University
Other Study IDs: Cancer survivor syndrome
Record Dates: First submitted 2023-03-10; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Cancer Survivors
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Myloid group: Patients diagnosed as Multiple Myeloma, treated, and not in relapse
  Interventions: Other: questionnaire
- Lymphoid group: Patients diagnosed as having lymphoma, treated, and not in relapse
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — The symptom related checklist questionnaire, Quality of life questionnaire, Coping strategies questionnaire, Distress thermometer

SUMMARY:
General objective: to improve care for haematological cancer survivors. This study will (i) Estimate the incidence of cancer survivor syndrome (CSS) in adult Egyptian patients with haematological neoplasms (HN). (ii) Asses the risk factors of CSS in patients with HN. (iii) Study the effect of CSS on quality of life in patients with HN. (iv) To explore coping strategies of patients with HN having CSS

DETAILED DESCRIPTION:
According to the American Cancer Society the term cancer survivor refersto people who have no signs of cancer after finishing treatment, people receiving extended treatment over a longer period of time to control the cancer or reduce risk of its return, and people with advanced cancer. Most hematologic malignancies (HM) are incurable and typically follow unpredictable remitting-relapsing pathways associated with varying need for treatment, which may be distressing for patients. Distress symptoms and psychological disorders secondary to cancer have also been shown to have significant negative consequences for both the patient and the family.

Maladaptive coping and abnormal illness behavior have been associated with psychiatric conditions, with negative effects on adherence to treatment, health behavior, and quality of life (Grassi et al 2017). Moreover, an increased length of stay in the hospital and/or an increased time in rehabilitation have been found to be more common among patients showing psychiatric symptoms, especially depression, than those with normal adjustment to illness (Cordova et al 2017). Unfortunately, cancer-related distress is commonly underrecognized and subsequently undertreated especially for patients with HM in developing countries. Search in literature revealed several screening methods for the psychological consequences of cancer such as Distress Thermometer , Symptom related checklist questionnaire, Quality of life questionnaire, Coping strategies questionnaire. Also, guidelines for the management of psychological distress have been developed by several scientific cancer associations.

ELIGIBILITY:
Inclusion Criteria:

* a. Inclusion criteria:

  1. Age will be more than or equal 18 years old regardless with six.
  2. Patients have been clinically diagnosed with haematological cancers.
  3. Being Native Egyptian patients.

Exclusion Criteria:

* History of psychiatric disorders. b) Having other concomitant haematological diseases or solid neoplasm or relapse or other chronic disorders

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Cancer survivor syndrome patients with haematological malignancy divided into two groups:
  Group 1: Myeloid neoplasms. Group 2: Lymphoid neoplasms in remission. The questionnaires will be collected from January 2023 to January 2025 in the Department of Hematology from Assiut University Hospital. This study will be approved from the Committee on Human Experimentation of Assiut University
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of cancer survivor syndrome (CSS) | 2 years
  Estimate the incidence of cancer survivor syndrome (CSS) in adult Egyptian patients with hematological neoplasm neoplasms (HN)

SECONDARY OUTCOMES:
Asses the risk factors of CSS | 2 years
  Asses the risk factors of CSS in adult Egyptian patients with hematological neoplasm neoplasms (HN)
Study the effect of CSS on quality of life | 2 years
  Study the effect of CSS on quality of life in adult Egyptian patients with hematological neoplasm neoplasms (HN)
Exploring coping strategies | 2 years
  To explore coping strategies of adult Egyptian patients with hematological neoplasm neoplasms (HN) in CSS.

CONTACTS AND LOCATIONS:
Overall Officials: Safaa AA Khaled, MD, PhD, Study Director — Professor, Department of Internal Medicine, Assiut University; Zain E Ahmed, MD, PhD, Study Chair — Professor, Department of Internal Medicine, Assiut University; Roaa M Saleh, MD, Principal Investigator — Resident Doctor, Department of Internal Medicine, Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hann D, Winter K, Jacobsen P. Measurement of depressive symptoms in cancer patients: evaluation of the Center for Epidemiological Studies Depression Scale (CES-D). J Psychosom Res. 1999 May;46(5):437-43. doi: 10.1016/s0022-3999(99)00004-5. PMID 10404478
- [Background] Albrecht TA, Rosenzweig M. Management of Cancer Related Distress in Patients with a Hematological Malignancy. J Hosp Palliat Nurs. 2012 Oct 1;14(7):462-468. doi: 10.1097/NJH.0b013e318268d04e. PMID 23002383
- [Background] Grassi L, Spiegel D, Riba M. Advancing psychosocial care in cancer patients. F1000Res. 2017 Dec 4;6:2083. doi: 10.12688/f1000research.11902.1. eCollection 2017. PMID 29259774